CLINICAL TRIAL: NCT01418846
Title: Determination of Voriconazole Levels in Saliva - Validation in Specific Subsets of Patients.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML7401
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2013-02

CONDITIONS: Pneumology; Hematology; Internal Medicine; Pediatrics
Keywords: voriconazole; saliva; pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- adult hematology patients
- pediatric patients age 5-18years
- adult pneumology patients

SUMMARY:
The purpose of this study is to investigate the intra-saliva penetration of voriconazole in different subpopulations. The goal is to develop, optimize and validate an easy, non-invasive and painless procedure for Therapeutic Drud Monitoring of voriconazole that can be used in children, ambulatory patients and in patients in whom blood drawing is difficult.

ELIGIBILITY:
Inclusion Criteria:

* patients from the adult hematology ward treated with voriconazole
* pediatric patients treated with voriconazole, age 5-18 years
* patients from the pneumology ward treated with voriconazole

Exclusion Criteria:

* Age under 5 years
* Women who are pregnant or lactating
* Mucositis stage 3 or 4 (WHO)
* Patients which received the following drugs within 14 days before study entry: rifampicin, rifabutin, carbamazepine, phenytoin, phenobarbital, nevirapine, efavirenz and barbiturates.
* Patients which received the following drugs within 24hours before study entry: quinidine, ergotamine, sirolimus, saquinavir, amprenavir, nelfinavir, ritonavir and sulphonylureas.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at the pneumology ward, adult hematology ward and all hospitalized pediatric patients, treated with voriconazole.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Voriconazole pharmacokinetics in saliva and plasma in different patient populations | One day at steady state of voriconazole plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Kim Vanstraelen, R.Ph., Principal Investigator — Catholic University of Leuven, Faculty of Pharmacy, division Hospital Pharmacy
Locations (3):
- Belgium (3):
  - University Hospital Brussels - Cystic Fibrosis Clinic, Brussels, Brussels Capital
  - Ghent University Hospital - Cystic Fibrosis Clinic, Ghent, East Flanders
  - University Hospitals Leuven, Leuven, Vlaams-Brabant